CLINICAL TRIAL: NCT03009903
Title: Evaluation and Detection of Facial Propionibacterium Acnes Bacteria and Phage Using Pore Strips in Humans
Brief Title: Evaluation and Detection of Facial Propionibacterium Acnes Bacteria and Phage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MBcure Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MBC-CL-01-2016
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- P. acne subjects: 14-50 year of age, P. acne diagnosed subjects
- None P. acne subjects: 14-50 year of age, none P. acne diagnosed subjects

SUMMARY:
This multi-center, outpatient study will extract and evaluate the presence of facial P. acnes bacteria and phage strains using pore strips on up to 400 human subjects.

DETAILED DESCRIPTION:
This multi-center, outpatient study will extract and evaluate the presence of facial P. acnes bacteria and phage strains using pore strips on up to 400 human subjects. An additional P. acnes visual detection method (VISIOPOR ® PP34N) will be used in this study as per PI decision to explore whether there is a correlation between P. acnes bacterial presence and fluorescent signal.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 14 to 50 years of age inclusive at the time of signing the informed consent
2. Able to provide written informed consent
3. Subjects who are willing to undergo pore strip treatment using the cosmetically acceptable pore strip product
4. Subjects who are willing to provide comprehensive demographic data using questionnaires

Exclusion Criteria:

1. Unwilling or unable to follow the procedures outlined in the protocol
2. Subjects treated with isotretinoin or tretinion during the 6 months prior to visit 1
3. Subjects treated with immunosuppressant agents
4. Pregnant subjects

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be male or female, ages 14-50. Healthy subjects and acne diagnosed subjects.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Detection and analysis of facial P. acnes presence | Day 0 and week 8 (optional)

SECONDARY OUTCOMES:
Assessing correlation between phage and P. acnes using: a. Demographic Questionnaire b. Visual Supportive Methodology (VISIOPOR ® PP34N) as per PI decision. | Day 0 and week 8 (optional

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shapiro, MD, Principal Investigator — Maccabi Healthcare Services, Israel

IPD SHARING:
Plan to Share IPD: No
2 sites to be activated. Dr. Shapiro is considered as PI in both sites